CLINICAL TRIAL: NCT04359264
Title: Direct Income SupporT and Advice Negating Spread of Epidemic COVID-19: a Randomized Controlled Trial (DISTANSE COVID-19 RCT)
Brief Title: Direct Income SupporT and Advice Negating Spread of Epidemic COVID-19: a Randomized Controlled Trial
Acronym: DISTANSE COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-081
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cash transfer (Experimental)
  Interventions: Other: Cash transfer
- Control (No Intervention)

INTERVENTIONS:
Other: Cash transfer — Cash transfer of $1000
  Arms: Cash transfer

SUMMARY:
This is a clinical trial of a cash transfer on symptoms consistent with COVID-19 and adherence to physical distancing guidance.

ELIGIBILITY:
Inclusion Criteria:

* trouble "making ends meet at the end of the month" due to COVID-19 related disruptions

Exclusion Criteria:

* confirmed positive for COVID-19 based on laboratory testing
* current symptoms consistent with COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Symptoms consisent with COVID-19 | 14 days
  32-item Influenza Patient-reported Outcome (FLU-PRO) symptom score. Higher score is worse.

SECONDARY OUTCOMES:
Number of close contacts | Sum of contacts on days 5, 10 and 14
Number of participants with positive test for COVID-19 | 14 days
Self-reported health based on the single question: "In general, would you say your health is.." | 14 days
Ability to make ends meet based on the single question: "At the end of the month, are you able to make ends meet?" | 14 days

OTHER OUTCOMES:
Health care utilization | 14 days
Food security | 14 days
  Three-items (worry about food running out, food did not last, balanced meals)
Cost-related medicine non-adherence | 14 days
  Single item: "During the last two weeks, did you or any member of your household not take a medication, skip some doses, split pills or do anything else to make a medication last longer due to the cost?"

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Municipality of Assiginack Family Health Team, Assiginack, Ontario
  - St Michael's Hospital Academic Family Health Team, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Persaud N, Thorpe KE, Bedard M, Hwang SW, Pinto A, Juni P, da Costa BR; DISTANSE COVID-19 (Direct Income SupporT and Advice Negating Spread of Epidemic COVID-19: a randomized controlled trial) study team. Cash transfer during the COVID-19 pandemic: a multicentre, randomised controlled trial. Fam Med Community Health. 2021 Dec;9(4):e001452. doi: 10.1136/fmch-2021-001452. PMID 34924360